CLINICAL TRIAL: NCT01372787
Title: Quality of Life and Care Needs in Patients With Persistent or Recurrent Platinum-Resistant Ovarian, Fallopian Tube, and Peritoneal Cancer
Brief Title: Quality of Life and Care Needs of Patients With Persistent or Recurrent Ovarian Cancer, Fallopian Tube Cancer, or Peritoneal Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Other Study IDs: GOG-0267; NCI-2011-02547 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000701477; GOG-0267 (Other: NRG Oncology); GOG-0267 (Other: DCP); GOG-0267 (Other: CTEP); U10CA101165 (NIH)
Record Dates: First submitted 2011-06-11; First posted 2011-06-14 (Estimated); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Anxiety; Fatigue; Nausea and Vomiting; Neurotoxicity Syndrome; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma; Stage I Ovarian Cancer AJCC v6 and v7; Stage IA Fallopian Tube Cancer AJCC v6 and v7; Stage IB Fallopian Tube Cancer AJCC v6 and v7; Stage IC Fallopian Tube Cancer AJCC v6 and v7; Stage II Ovarian Cancer AJCC v6 and v7; Stage IIA Fallopian Tube Cancer AJCC v6 and v7; Stage IIB Fallopian Tube Cancer AJCC v6 and v7; Stage IIC Fallopian Tube Cancer AJCC v6 and v7; Stage III Ovarian Cancer AJCC v6 and v7; Stage III Primary Peritoneal Cancer AJCC v7; Stage IIIA Fallopian Tube Cancer AJCC v7; Stage IIIB Fallopian Tube Cancer AJCC v7; Stage IIIC Fallopian Tube Cancer AJCC v7; Stage IV Fallopian Tube Cancer AJCC v6 and v7; Stage IV Ovarian Cancer AJCC v6 and v7; Stage IV Primary Peritoneal Cancer AJCC v7
MeSH Terms: conditions — Anxiety Disorders; Fatigue; Nausea; Vomiting; Neurotoxicity Syndromes; Fallopian Tube Neoplasms; Ovarian Neoplasms

GROUPS / COHORTS (1):
- Arm I
  Interventions: Procedure: Assessment of Therapy Complications; Other: Medical Chart Review; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Assessment of Therapy Complications — Ancillary studies
Other: Medical Chart Review — Ancillary studies
  Other Names: Chart Review
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial studies the quality of life and care needs of patients with persistent or recurrent ovarian cancer, fallopian tube cancer, or peritoneal cancer. Studying quality of life in patients with cancer may help determine the effects of gynecologic cancer and may help improve the quality of life for future cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the prevalence and severity of patient-reported symptoms in patients with platinum-resistant ovarian, fallopian tube, and peritoneal cancers at study entry and at three and six months post-enrollment.

SECONDARY OBJECTIVES:

I. To explore the unmet needs of these women at study entry and at three and six months post-enrollment (Exploratory) II. To explore the overall quality-of-life (QOL) of these women at study entry and at three and six months post enrollment. (Exploratory) III. To explore the relationship between patient-reported symptoms and overall QOL, current cancer therapy (yes/no), and treatment responses (if on cancer therapy). (Exploratory)

OUTLINE: This is a multicenter study.

Patients complete the Needs at the End-of-Life Screening Tool (NEST), the Functional Assessment of Cancer Therapy ? Ovarian (FACT-O), the FACIT-Fatigue Subscale (FACIT-F), the National Comprehensive Cancer Network (NCCN) FACT Ovarian Symptom Index-18 (NFOSI-18), the FACT/GOG-AD subscale for ovarian cancer-related abdominal discomfort, and the FACT/GOG-Neurotoxicity (FACT/GOG-NTX) Scale quality-of-life questionnaires at baseline and at 3 and 6 months during office or clinic visits or via telephone or mail. Patients' demographic and therapy information, such as current age, ethnicity, marital status, employment status, prior chemotherapy regimens/cancer treatment, disease status (if available), performance status, patient care information, and current cancer therapy are also collected.

After completion of study participation, patients are followed up every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with persistent or recurrent epithelial ovarian cancer, peritoneal cancer, or fallopian tube cancer

  * Platinum-resistant (less than 6 months from date of last platinum therapy to date of first evidence of recurrent or persistent disease) disease as measured by any of the following:

    * Imaging
    * Physical exam
    * CA-125 that is twice the upper limit of normal on two occasions with at least one week apart
  * No patients who have platinum resistant or refractory disease after more than 6 months since prior therapy
* Criteria for patients on cancer therapy (e.g., chemotherapy, non-cytotoxic regimens, hormone therapy, or radiation therapy) include recurrent or persistent disease defined as having measurable disease per RECIST (Version 1.1)

  * Patients not on chemotherapy are also eligible and are not required to have RECIST criteria
* Life expectancy of at least 6 months
* Patients with any performance status, yet with the ability to verbally consent and participate in the first assessment

  * Study measures will be administered in the office/clinic setting, or for study participants who are unable to attend clinics, via telephone or mail (telephone is the preferred back-up means)
* Patients may have or have had a prior non-gynecologic malignancy within 5 years prior to study enrollment; however, they must have completed all treatments for the disease and have no evidence of disease at the time of enrollment, and ovarian, peritoneal, or fallopian tube cancer must be the primary life-threatening diagnosis
* Patient must be able to read and write English
* No patients receiving chemotherapy for platinum-sensitive ovarian cancer, peritoneal, or fallopian tube cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Sampling Method: Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2011-04-12 (Actual); Primary Completion 2014-01-31 (Actual)

PRIMARY OUTCOMES:
Prevalence and severity of patient-reported symptoms as measured by the NFOSI-18, the FACIT-F subscale, and the FACT/GOG-AD and NTX subscales | Up to 6 months
  Assessed at baseline, and at 3 and 6 months. The prevalence of a patient-reported symptom will be determined by the percentage of living patients reporting the presence of a symptom at the assessment time point.

CONTACTS AND LOCATIONS:
Overall Officials: Vivian E von Gruenigen, Principal Investigator — NRG Oncology
Locations (144):
- United States (144):
  - University of Colorado Hospital, Aurora, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Sudarshan K Sharma MD Limited-Gynecologic Oncology, Hinsdale, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - McFarland Clinic PC - Ames, Ames, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - Maine Medical Center-Bramhall Campus, Portland, Maine
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Massachusetts Memorial Health Care, Worcester, Massachusetts
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Beaumont Hospital ? Dearborn, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Saint Dominic-Jackson Memorial Hospital, Jackson, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Morristown Medical Center, Morristown, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Cleveland Clinic Akron General, Akron, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Main Line Health NCORP, Wynnewood, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Chattanooga's Program in Women's Oncology, Chattanooga, Tennessee
  - Memorial Hermann Texas Medical Center, Houston, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin